CLINICAL TRIAL: NCT00004043
Title: Phase II Study of Pulse Calcitriol in Patients With Rising PSA After Definitive Treatment for Prostate Cancer
Brief Title: Calcitriol in Treating Patients With a Rising PSA Level Following Treatment for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067041; OHSU-5231; OCC-HOR-98068-L; NCI-V99-1542
Record Dates: First submitted 1999-12-10; First posted 2004-06-17 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: calcitriol

SUMMARY:
RATIONALE: Calcitriol, a form of vitamin D, may be able to prevent or slow the growth of prostate cancer cells.

PURPOSE: Phase II trial to study the effectiveness of calcitriol in treating patients who have a rising PSA level following previous treatment for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response to pulse calcitriol in patients with previously treated adenocarcinoma of the prostate with rising PSA levels. II. Assess the impact of this regimen on the slope of the PSA rise in these patients. III. Determine the qualitative and quantitative toxic effects of this regimen in these patients. IV. Assess the impact of this regimen on the quality of life of these patients.

OUTLINE: All patients remain on a reduced calcium diet for the duration of the study. Twelve hours prior to treatment, patients begin drinking 4-6 glasses of extra fluid for 3 days. Patients receive oral calcitriol over 4 hours weekly. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, every 4 weeks during treatment, and at the end of the study. Patients are followed for at least 1 month.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven adenocarcinoma of the prostate previously treated with prostatectomy or definitive radiotherapy Rising PSA after post definitive therapy nadir on at least 3 measurements at least 2 weeks apart PSA at least 0.4 ng/mL for prostatectomy patients PSA at least 1.0 ng/mL for radiotherapy patients

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 2 months Hematopoietic: Not specified Hepatic: Not specified Renal: Phosphate no greater than 4.2 mg/dL Creatinine no greater than 1.3 mg/dL Calcium no greater than 10.5 mg/dL No history of hypercalcemia Cardiovascular: No significant heart disease No myocardial infarction within past 3 months No history of heart failure Cardiac ejection fraction at least 30% Other: No other significant active medical illness that would preclude compliance Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior systemic chemotherapy for metastatic prostate cancer (except neoadjuvant treatment for localized prostate cancer) Endocrine therapy: No prior systemic hormonal therapy for prostate cancer (except neoadjuvant treatment for localized prostate cancer) Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: No other concurrent systemic therapy for metastatic prostate cancer At least 30 days since other prior investigational drugs No concurrent digoxin At least 7 days since prior thiazide diuretic therapy No concurrent magnesium containing antacids, bile resin binding drugs, or calcium supplements

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-02; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Beer, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Result] Lowe BA, Henner WD, Lemmon DD, et al.: Long term administration of high dose weekly oral calcitriol in patients with a rising PSA after definitive treatment for prostate cancer (PC): a phase II study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-2446, 2002.